CLINICAL TRIAL: NCT07260968
Title: Facilitating Lactation Through Optimized Workflows - Evaluating the Efficiency of Pumping Protocols and Cellular Mechanisms of Milk Production
Acronym: FLOW
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Cornell University (Other)
Responsible Party: Principal Investigator, Casey Rosen-Carole, MD, MPH, MSEd, NABBLM-C, FABM, University of Rochester
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00011127
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Low Milk Supply

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pumping 6-8 times a day (also known as triple-feeding protocol) (Experimental)
  Interventions: Other: Pumping frequency intervention
- Pumping 3-4 times a day (lower frequency of pumping) (Experimental)
  Interventions: Other: Pumping frequency intervention
- No additional pumping will be recommended (mothers can choose to pump as they desire) (Experimental)
  Interventions: Other: Pumping frequency intervention

INTERVENTIONS:
Other: Pumping frequency intervention — In this randomized clinical trial, we will evaluate whether a lower frequency of pumping (3-4 times/day) or no additional pumping recommendations can lead to higher compliance, an increase in milk production, and a longer duration of breastfeeding.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of two different breast pumping protocols in increasing milk production among lactating individuals diagnosed with primary low milk supply, and to investigate the associated molecular, hormonal, and inflammatory mechanisms driving milk output.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Lactating parents of singleton, term infants less than 3 months of age
* Intend to breastfeed and are breastfeeding (at the breast) at least 3 times per day

Exclusion criteria:

* Twins and other multiples
* Contraindications to or unable to breastfeed
* Major congenital anomaly or unexpected surgery
* Elevated maternal depression
* Low milk transfer
* No electricity or smartphone access

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2027-12-20 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Milk Production | 6 month follow-up
  The study will measure milk production using a 24-hour test weighing (weighing infants before and after each feed) before and after the intervention.